CLINICAL TRIAL: NCT00212043
Title: Phase I/II Trial of Infusional Gemcitabine in Combination With Carboplatin in Chemonaive Non-small Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRG L08/99
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2008-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: randomised phase II trial gemcitabine and carboplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Gemcitabine

INTERVENTIONS:
Drug: carboplatin and gemcitabine

SUMMARY:
Hypothesis - Infusional gemcitabine may give better intracellular pharmacologic activation and be more effective clinically in non-small cell lung cancer

DETAILED DESCRIPTION:
Objectives of study:

1. to compare the response rate of carboplatin and constant rate infusion gemcitabine to the response rate of gemcitabine given in the standard 30-minute infusion
2. to compare the toxicity experience in both arms
3. To compare the time to progression in both study arms, and overall survival
4. To compare the quality of life on both study arms using the EORTC QLQ-C30 and QLQ-LC13.

   Inclusion criteria
   * Histologically or cytologically confirmed NSCLC.
   * Stage IIIB unsuitable for radical radiation (eg. with cytologically proven malignant effusion) or stage IV disease as defined by the AJCC criteria (see appendix 1).
   * Karnofsky performance status 70% or higher (see appendix 2).
   * Presence of at least one bidimensionally or unidimensionally measurable, non-CNS, indicator lesion defined by radiologic study or physical examination.
   * No previous chemotherapy for advanced disease. Prior neoadjuvant or adjuvant chemotherapy, or chemotherapy given concurrently with radiotherapy for non-metastatic disease, is allowed if the last dose was given 6 months or more before study entry.
   * Patients with recurrent disease after primary surgery and/or radiotherapy will be eligible.
   * For patients with previous radiotherapy, the indicator lesion(s) must not be within previous radiation field. The last dose of radiotherapy should be at least 3 weeks prior to study entry. The total radiotherapy received should not be more than 30% of the bone marrow.
   * Screening laboratory criteria:

   WBC count > 3500/microl Neutrophils > 2000/microl Platelet count > 100,000/microl Hemoglobin > 9 g/dl (transfusion allowed)

   Serum creatinine < 133 micromol/l, or Creatinine clearance > 30 ml/min, based on the Cockcroft formula (see section 5.1.1)

   Bilirubin < 1.5 x upper limit of normal ALT/AST < 2 x upper limit of normal if liver metastases are absent < 5 x upper limit of normal if liver metastases are present
   * Aged 18 years and above.
   * Life expectancy > 3 months.
   * Written informed consent.

   4.2 Exclusion criteria

   The following conditions will render patients ineligible to participate in this study:
   * Patients with only evaluable disease.
   * Active uncontrolled infection.
   * Pregnant or lactating women.
   * Females of childbearing potential who are unwilling to avoid pregnancy, for the duration of the study.
   * Presence of any underlying medical conditions which in the investigators opinion would make the patient unsuitable for treatment.
   * Concomitant malignancies or previous malignancies other than NSCLC within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin, carcinoma-in-situ of the cervix, or stage A low grade prostate cancer.
   * Patients with CNS and/or leptomeningeal metastases; unless asymptomatic and not receiving corticosteriod therapy.

   4.3 Inclusion and exclusion criteria for phase I patients

   The exclusion criteria are the same as above.

   The inclusion criteria are the same as above except for the following groups of patients, which are allowed in the phase I study:
   * Patients with evaluable disease only (with no measurable lesions).
   * Patients with one (and only one) line of chemotherapy for advanced NSCLC, excluding patients who had received prior platinium and/or gemcitabine.
   * Patients with indicator lesions in previous radiation field.

   Measurability of indicator lesions
   * Measurable: The lesion can be measured accurately in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10mm with spiral CT scan.
   * Non-measurable: All other lesions including small lesions (longest diameter <20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly non-measurable lesions. Lesions considered to be truly non-measurable include the following: bone lesions, leptomeningeal disease, ascites, pleural/cutis/pulmonis, abdominal masses that are not confirmed and followed by imaging techniques, and cystic lesions.
   * Target Lesions: All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total representative of all involved organs should be identified as target lesions and be recorded and measured at baseline. Target lesions should be selected on the basis of their size (lesion with the longest diameter) and their suitability for accurate measurements (either by imaging techniques or clinically). A sum of the longest diameter (LD) for all target lesions will be calculated and reported as the baseline sum LD. The baseline sum LD is used as the reference by which to characterize the objective tumor response. If there are > 10 measurable lesions, those not selected as target lesions will be considered together with non-measurable disease as non-target lesions.
   * Non-target Lesions: All non-measurable lesions (or sites of disease) plus any measurable lesions over and above the 10 listed as target lesions. Measurements are not required but these lesions should be noted at baseline and should be followed as "present" or "absent".
   * Any tumour measurement relying solely on physical examination should be verified by a second physician.
   * The same diagnostic imaging method must be used throughout the study to evaluate the lesions.
5. TREATMENT PLAN

   5.1 Phase I study

   5.1.1 Carboplatin

   The starting dose of carboplatin is given at a fixed dose at a target AUC of 5 over 1 hour on day 1 in both arms of the study. Carboplatin will be given before gemcitabine in all patients. The dose is repeated every 21 days and will be calculated using the Calvert formula:

   Dose of carboplatin (mg) = [calculated glomerular filtration rate (GFR) + 25] x 5

   The GFR will be calculated according to the Cockroft-Gault formula:

   GFR (ml/min) = (140 - age) x body weight (in kg) / 0.81 x serum creatinine (micromol/l)

   For female, the correction factor is 0.85 (x calculated GFR)

   5.1.2 Infusional gemcitabine

   Infusional gemcitabine is given at a constant rate of 10 mg/m2 per minute in all patients on days 1 and 8, the cycle is repeated every 21 days. Dose escalation is achieved by increasing the duration of infusion. The total dose of gemcitabine is re-constituted in 500 ml of normal saline and infused through a peripheral or central venous line.

   5.2.1 Treatment courses

   Prior to initiating treatment, eligible patients will be randomised to receive gemcitabine given either in the standard short 30 minutes infusion, or constant rate prolonged infusion over the duration determined in the phase I study. All patients in both arms will receive carboplatin at a dose of AUC of 5 over 1 hour.

   Standard arm

   Carboplatin AUC of 5 over 1 hour, day 1, followed by Gemcitabine 1000 mg/m2 over 30 min, day 1 and 8 Cycle is repeated every 21 days

   Study arm

   Carboplatin AUC of 5 over 1 hour, day 1, followed by Gemcitabine 10 mg/m2/min at MTD, day 1 and 8 Cycle is repeated every 21 days

   Supportive treatment
   * All patients should receive pre-medications to prevent nausea and vomiting according to local policy.
   * No prophylactic growth factors are allowed.
   * Growth factor is allowed only in the rescue setting, eg. prolonged grade 4 neutropenia for more than 7 days, or for febrile neutropenia.

   5.2.2 Dosing in cycle 2 and subsequent cycles

   The next treatment cycle will begin on schedule providing

   • There is no evidence of tumour progression
   * Neutrophils ~ 2 x 109/L
   * Platelets ~ 100,000 x 109/l
   * Absence of grade 2 or above non-haematological toxicity

   5.2.3 Dose modifications

   5.2.3.1 General rules
   * No intra-patient dose escalation is allowed.
   * Any patient who requires a dose reduction will not be eligible for any dose escalation for the remainder of the study.
   * Treatment may be delayed up to day 35 to allow a patient sufficient time for recovery from treatment related toxicity. Any patient who cannot proceed to the next cycle by day 35 will be discontinued from the study.

   5.2.3.2 Dose modifications based on haematologic toxicity

   Adjustment based on day 8 count Platelets (x 109/l) ANC (x 109/l) Action > 75 and > 1.0 Proceed with day 8 dose > 75 and 0.5 - 1.0 Proceed with reduced dose 50 - 75 and ~ 0.5 Proceed with reduced dose < 50 and/or < 0.5 Omit dose When day 8 dose is reduced, the same reduced dose will be used for the following cycle.

   When day 8 dose is omitted, the cycle is completed, and the next cycle will be scheduled on day 22, with dose reduction.

   Dose adjustment based on nadir count Platelets (x 109/l) ANC (x 109/l) Action ~ 25 with no bleeding and ~ 0.5 or < 0.5 for < 7 days No change < 25 or < 50 with bleeding and/or < 0.5 for > 7 days Dose reduction (see below) Any and < 0.5 and fever Dose reduction Recurrence of any of the above after 2 dose reductions Off study

   Adjustment based on day 22 count Platelets (x 109/l) ANC (x 109/l) Action

   ~ 100 and > 2.0 Proceed with next cycle < 100 and/or < 2.0 Delay 1 week Maximum delay of 2 weeks (next cycle must start by day 35 to remain on study)

   Dose reduction schema First Reduction Second reduction Third reduction Carboplatin AUC 4.5 AUC 4.0 Off study Gemcitabine (standard arm) 750 mg/m2 (1000 mg/m2 x 75%) 500 mg/m2 (1000 mg/m2 x 50%) Off study Infusional Gemcitabine 75% of Phase II duration 50% of previous infusion duration Off study

   5.2.3.3 Dose modifications for non-haematologic toxicity

   Any grade 3 or 4 non-haematologic toxicity, except for nausea and vomiting and fatigue and reversible transaminitis, will render patient off study.

   Non-haematologic toxicity must be less than grade 2 before proceeding to the next cycle. If they are higher than grade 2, treatment is delayed for 1 week. Treatment may be delayed for a maximum of 2 weeks.

   5.2.4 Treatment duration

   Responding patients will receive up to six cycles of chemotherapy.

   After treatment completion or withdrawal, patients may continue to receive further treatment at the discretion of their physician.

   Screening evaluations

   The following screening investigations must be performed within 28 days of day 1 of cycle 1:
   * Complete staging and documentation of tumour status - baseline chest x-ray, CT thorax, abdomen, brain and bone scan if clinically indicated.

   The following screening evaluations and investigations must be performed within 14 days of the first dose of therapy and includes the following:

   • Consent

   • Complete medical history, include details of symptoms, prior treatments, any residual toxicity, concomitant medical conditions and medications

   • Physical examinations, including documentation of all palpable lesions, vital signs, body weight and height, and KPS.

   • Documentation of indicator lesion(s) to include date of assessment, description of lesion site, dimensions, and type of diagnostic study to follow lesion. The same diagnostic method must be used throughout the study to evaluate a lesion.

   The following tests must be performed within 7 days of the first dose of therapy and includes the following:
   * Full blood count
   * Serum electrolytes and liver enzymes, total calcium and magnesium
   * Serum pregnancy test, if applicable
   * Dipstick urinalysis - if dipstick is positive for protein or blood, a complete microscopic examination is required

   8.3 Evaluation during treatment

   Prior to day 1 of each cycle

   • History and physical examination

   • Assess and record toxicities from prior course. Assign appropriate toxicity grades (see Appendix 4).

   • Record all medications taken since the last cycle.

   • Weight measurement for re-calculation of body surface area and creatinine clearance

   • Assessment of symptoms of disease (QoL questionnaire should be given and filled by patient before assessment by investigator).
   * Assessment of performance status
   * Full blood count, electrolytes and liver enzymes (if day15 levels are abnormal).
   * Urine dipstick analysis, if the baseline result is abnormal
   * Clinical tumour measurements should be obtained prior to every cycle of treatment
   * Radiographic tumour measurements should be obtained after every 2 cycles of treatment.
   * Modify dose of the next cycle if necessary (see section 5.2.3).

   Day 8 assessment

   • Full blood count

   Day 15 assessment

   • Full blood count, electrolytes and liver enzymes

   8.4 Evaluation of response

   Patients will be evaluable for response after 2 cycles of therapy. Clinical tumour measurements should be performed prior to every cycle of treatment. Radiographic tumour measurements should be obtained after every 2 cycles of treatment.

   If a patient meets the response criteria (see section 7) for CR, PR or SD for the first time, another clinical and radiographic tumour assessment will be performed 4 or more weeks later to document that the response has lasted at least 4 weeks.

   Clinical tumour assessment after every cycle and radiographic tumour response after every 2 cycles will continue until completion of treatment or patient withdrawal.

   8.5 Post-treatment follow-up

   Responding patients will be reviewed every 2 monthly after completion of chemotherapy. Clinical tumour assessment will be carried out 2 monthly. Radiographic tumour assessment will be done every 4 monthly. These will continue until disease progression is documented.

   Patients who never had a response, and patients with disease progression after a previously documented response will be followed every 3 monthly for survival data.

9. TREATMENT COMPLETION AND WITHDRAWAL

A patient will be considered as completing the treatment if:

* Patient has completed 6 cycles of therapy.
* Patient has a confirmed CR or confirmed PR and received at least 4 cycles of therapy and the investigator does not feel further therapy is indicated.
* Patient maintained a status SD for at least 8 weeks on treatment and received at least 2 cycles of treatment.
* Patient has PD after completing at least one full course of treatment.
* A patient is removed from the study due to unacceptable toxicity.

Patients may be withdrawn from the treatment for the following reasons:

* Adverse experience, including intercurrent illness or unacceptable toxicity.
* If attending physician thinks a change of therapy would be in the best interest of the patient.
* Protocol violation (including non-compliance).
* Patient withdrawal at his/her request, for reasons other than those above.
* Lost to follow-up.

All patients will be followed for status of disease and survival until death. 10. QUALITY OF LIFE (QoL) ASSESSMENT

It is essential to explain to the patient that the QoL assessment is an important part of the trial, and that all sections should be answered even if the patient feels them to be irrelevant. It should be emphasized that the completion of these forms helps doctors find out more about the effects of treatment on patients' well-being.

A named contact person other than the responsible clinician managing the patient in the context of the trial, must be appointed to take responsibility for the administration, collection and checking of the completed EORTC QLQ-C30 and QLQ-LC13 questionnaire. The questionnaire must be taken before consultation with the clinician, according to the EORTC guidelines for QoL assessment. They should be checked to ensure that all questions have been answered; if necessary go back to the patient immediately and ask him or her to fill in any missing items. If an assessment is missed because of administrative failure, the patient should be contacted by telephone or letter and an arrangement should be made for the questionnaire to be taken within a week of the scheduled assessment.

The questionnaire may be filled in by the patient if he/she is able to read and understand the language of the questionnaire. Otherwise, the named person for administering the QoL should read out the questions as written, in the language the patient understands, and record the response to each question without prejudicing his/her answer. The mode of delivery should be noted in the questionnaire.

11. RANDOMISATION PROCEDURE

Study participants will be randomly assigned to receive either gemcitabine given in the conventional 30 minutes infusion, or protracted infusion, both in combination with carboplatin.

11.1 Stratification

Stratified randomization will be carried out using the minimization method based on the following factors:

(i) Centre (National University Hospital, Sydney Cancer Centre, Johns Hopkins-NUH International Medical Centre) (ii) Karnofsky performance status (90 - 100% vs 70 - 80%) (iii) Stage of disease (IIIB vs IV)

11.2 Registration

Patients will be entered into the trial by a telephone call to the National Medical Research Council (NMRC) Clinical Trials & Epidemiology Research Unit (CTERU), Singapore (+65 220-1292) between 0830 to 1730 hours Monday to Friday, and 0830 to 1230 hours Saturday (Singapore time), or by Fax (+65 220-1485), stating that the patient is to be entered into the CTRG L08 or SQLU02 trial.

Informed written consent for entry into the study should be obtained prior to randomization. All eligibility criteria and consent form will be checked, and the stratification factors stated before treatment is allocated. The patient will be randomized to long infusional gemcitabine (L) or 30- minute short infusion gemcitabine (S), and allocated a trial number. The design will involve equal allocation of patients to the two treatments. Confirmation fax will be sent to the investigator.

12. STATISTICAL CONSIDERATIONS

The sample size calculation is carried out based on the statistical selection theory criterion as detailed in Simon et al (62) and Gibbons et al (63). Assuming a 90% probability of correctly selecting the best treatment, and anticipating a baseline response rate of 40%, then to detect a 15% superiority of the best treatment over the other, a trial size of 37 patients per treatment arm would be required. The total accrual target would thus be 74 patients.

13. STATISTICAL ANALYSES

Statistical analysis of all study endpoints will be carried out on an intention-to-treat basis. In the event of lost to follow-up, patients will still be included in the analysis for the duration that they are observed. The inherent comparability of results in this randomized phase II design using the statistical selection theory assures that the two treatments can be reliably ranked when large differences are obtained.

The best response will be used in the analysis of objective tumour response. In the case of adverse event, where multiple events of the same kind has occurred in a patient, only the maximum grade will be documented for the analysis. The tumour response rates and toxicities between treatment groups will be compared descriptively using estimates of proportions.

The response duration and time to response for responding patients will be assessed using appropriate descriptive statistics. The evaluation of progression-free and overall survival will be carried out using the Kaplan-Meier technique at 1-year follow-up. In the case of progression-free survival, patients whose disease has not progressed will be censored at the date last known to be alive. Similarly, the analysis of overall survival censors patients who are lost to follow-up or who remained alive at the date last known to be alive.

For each QoL dimension, changes in scores over time will be compared between treatment arms by means of appropriate graphical representation or descriptive statistics.

No interim analysis is planned for this randomised phase II trial.

14. ETHICAL CONSIDERATIONS

14.1 IRB/Ethics committee

Before study initiation, the protocol will be submitted for review and approval by the hospital and Ministry of Health research and ethics committee or equivalent group. Approval of the protocol and informed consent must be obtained.

14.2 Patient information

The responsible physician will inform the patient about the background and current knowledge of the treatment under study with special reference to known activity and toxicity. The patient will be told about the investigative nature of this treatment and in particular, the randomization process involved in this study. The patient will be told of his or her right to withdraw from the study at any time without any penalty with regards to the continuation of care at this institution and by the same physicians as he chooses. Before accrual, all patients will sign a written, informed consent form.

14.3 Informed consent

Informed consent should meet the requirement of the latest revision of the Declaration of Helsinki and any applicable regulations and guidelines such as the Good Clinical Practice (Singapore).

The study will be completely explained to each prospective candidate and the subject must give consent by signing and dating the consent form.

Consent must be obtained before any protocol-required procedures are performed, including any procedures not part of normal patient care.

Plasma dFdC and dFdU levels

Ten millilitres of blood will be drawn at 0 hours (baseline), 10 minutes, 30 minutes, 10 minutes before the end of the infusion, and 30 minutes, 1 hour, 2 hours after the end of the infusion. The blood will be drawn into 10 ml tubes (green topped) containing heparin and 5 micromol tetrahydrouridine. The tubes are then centrifuged at 3300 rpm for 15 minutes and the supernatant plasma is then transferred to plain tubes (red topped) for immediate storage at -80oC. Samples will be labeled with the patient's name, ID number, date, exact time of sample and protocol number. A pharmacokinetic form will accompany the plasma samples to the Pharmacology laboratory in the Department of Pharmacology, National University of Singapore, c/o Prof Lee How Sung.

DFdC and dFdU levels in plasma will be measured using reverse phase HPLC, as described by Grunewald (22). Briefly, 20 microl to 50 microl of plasma is injected onto a C18 mBondapak analytical column (Waters Associates, Inc.). Components will be separated with a mobile phase consisting of a 30 minute linear gradient starting with 100% solution A (0.5M ammonium acetate, pH = 6.8) and ending with 60% solution B (50% methanol in deionised water). Flow rate is at 1.5 ml/min. Detection wavelengths are 275 nm and 262 nm for dFdC and dFdU, respectively.

16.2 Intracellular dFdCTP levels

Samples of blood will be collected to assay intracellular dFdCTP. Only 3 samples per patient, obtained 10 minutes after the start and 10 minutes before the end of the infusion of gemcitabine, and one in the middle of infusion, will be assayed for dFdCTP.

Plasma is first separated from the blood by centrifugation at 3300 rpm for 20 minutes. Mononuclear cells are then isolated by Ficoll-Hypaque density gradient centrifugation and deoxyribonucleoside triphosphates are extracted with 0.4 NHClO4, and the acid-insoluble material is removed by centrifugation. The supernatant is then carefully neutralized to pH 7 with potassium hydroxide, and the precipitated KClO4 is then removed by centrifugation. An ion-exchange high performance liquid chromatography method is then used to separate and quantitate the dFdCTP.

17. STUDY ADMINISTRATION

17.1 Drug accountability

Stocks of gemcitabine will be supplied by Eli Lilly for trial purposes, and all these vials will be accounted for at the site pharmacy.

17.2 Maintenance of patients records

CTRG clinical report forms will be used to record data for this study. All patient clinical report forms will be faxed to the CTRG Office (+65 777-5545). A copy of each patients eligibility report form, randomization report form (for phase II), study schedule, consent forms, laboratory and radiological reports, and QoL assessment will be kept in the CTRG Office. All records will be kept for a period of 6 years following the date of study closure according to Singapore GCP guidelines

ELIGIBILITY:
Inclusion Criteria:

* • Histologically or cytologically confirmed NSCLC.

  * Stage IIIB unsuitable for radical radiation (eg. with cytologically proven malignant effusion) or stage IV disease as defined by the AJCC criteria (see appendix 1).
  * Karnofsky performance status 70% or higher (see appendix 2).
  * Presence of at least one bidimensionally or unidimensionally measurable, non-CNS, indicator lesion defined by radiologic study or physical examination.
  * No previous chemotherapy for advanced disease. Prior neoadjuvant or adjuvant chemotherapy, or chemotherapy given concurrently with radiotherapy for non-metastatic disease, is allowed if the last dose was given 6 months or more before study entry.
  * Patients with recurrent disease after primary surgery and/or radiotherapy will be eligible.
  * For patients with previous radiotherapy, the indicator lesion(s) must not be within previous radiation field. The last dose of radiotherapy should be at least 3 weeks prior to study entry. The total radiotherapy received should not be more than 30% of the bone marrow.
  * Screening laboratory criteria:

WBC count > 3500/microl Neutrophils > 2000/microl Platelet count > 100,000/microl Hemoglobin > 9 g/dl (transfusion allowed)

Serum creatinine < 133 micromol/l, or Creatinine clearance > 30 ml/min, based on the Cockcroft formula (see section 5.1.1)

Bilirubin < 1.5 x upper limit of normal ALT/AST < 2 x upper limit of normal if liver metastases are absent < 5 x upper limit of normal if liver metastases are present

* Aged 18 years and above.
* Life expectancy > 3 months.
* Written informed consent.

Exclusion Criteria:

* • Patients with only evaluable disease.

  * Active uncontrolled infection.
  * Pregnant or lactating women.
  * Females of childbearing potential who are unwilling to avoid pregnancy, for the duration of the study.
  * Presence of any underlying medical conditions which in the investigators opinion would make the patient unsuitable for treatment.
  * Concomitant malignancies or previous malignancies other than NSCLC within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin, carcinoma-in-situ of the cervix, or stage A low grade prostate cancer.
  * Patients with CNS and/or leptomeningeal metastases; unless asymptomatic and not receiving corticosteriod therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74
Dates: Start 2000-07; Study Completion 2004-02

CONTACTS AND LOCATIONS:
Overall Officials: Boon-Cher Goh, Study Chair — National University Hospital, Singapore

REFERENCES:
- [Derived] Tham LS, Wang LZ, Soo RA, Lee HS, Lee SC, Goh BC, Holford NH. Does saturable formation of gemcitabine triphosphate occur in patients? Cancer Chemother Pharmacol. 2008 Dec;63(1):55-64. doi: 10.1007/s00280-008-0707-9. Epub 2008 Feb 28. PMID 18305939